CLINICAL TRIAL: NCT00753597
Title: Immunotherapeutic Rescue of Steroidogenic Function in Autoimmune Adrenocortical Failure: Pilot Study
Brief Title: Rescue of Steroidogenic Capacity in Adrenocortical Failure Study (RADS)
Acronym: RADS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, SHS Pearce, Professor of Endocrinology, Newcastle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NUTH/2006/4071; EU ID: 2007-003062-18
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Autoimmune Adrenocortical Failure
Keywords: B cell depletion; steroidogenesis
MeSH Terms: interventions — Methylprednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receiving active treatment
  Interventions: Drug: Solu-medrone, Mabthera

INTERVENTIONS:
Drug: Solu-medrone, Mabthera — 125mg, 1gram, twice day 1 and day 15

SUMMARY:
This is a pilot study of B lymphocyte depletion therapy in an attempt to salvage adrenal steroidogenic capacity in ten subjects with early autoimmune Addison's disease. During the first twelve weeks of treatment, additional glucocorticoid therapy (prednisolone) will be given to ensure wellbeing and to rest the steroidogenic apparatus that is the target of the autoimmune attack. Glucocorticoids will be gradually withdrawn, in a controlled fashion, and adrenal function re-evaluated at 13, 26, 39 and 52 weeks. The primary endpoint will be restoration of steroidogenic function as judged by conventional endocrine indices of adrenocortical function. B cell depletion may ameliorate the autoimmune attack against adrenal cells, potentially allowing a state of immune tolerance to be restored with subsequent recovery of adrenal steroidogenic capacity.

ELIGIBILITY:
Inclusion Criteria:

* Clear evidence of primary adrenal failure (elevated ACTH, pigmentation, electrolyte disturbance)
* Basal or stimulated cortisol <400 nmol/l but >100nmol/l

Exclusion Criteria:

* Active viral infection, pregnancy or breast feeding, previous immunosuppression, diabetes, cardiorespiratory disease, renal failure, hepatic disease, cancer
* Calcified or enlarged adrenals on CT scan, active TB

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Peak serum cortisol, basal or post ACTH | 13, 26, 39, 52 weeks from first treatment

SECONDARY OUTCOMES:
21-OHase antibodies | 13, 26,39, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon Pearce, MD, FRCP, Principal Investigator — Newcastle University
Locations (1):
- Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Pearce SH, Mitchell AL, Bennett S, King P, Chandran S, Nag S, Chen S, Smith BR, Isaacs JD, Vaidya B. Adrenal steroidogenesis after B lymphocyte depletion therapy in new-onset Addison's disease. J Clin Endocrinol Metab. 2012 Oct;97(10):E1927-32. doi: 10.1210/jc.2012-1680. Epub 2012 Jul 5. PMID 22767640